CLINICAL TRIAL: NCT01855516
Title: Partial Thromboplastin Time After 72 Hours of Antithrombotic Prophylaxis Using Unfractionated Heparin: Comparison of a 2 Times Per Day Versus a 3 Times Per Day Dosage.
Brief Title: Partial Thromboplastin Time After 72 Hours of Antithrombotic Prophylaxis Using Unfractionated Heparin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NM2013-001
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Thrombosis
Keywords: Antithrombotic prophylaxis
MeSH Terms: conditions — Thrombosis | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UFH 5000 U three times a day (Active Comparator): Study subjects will be randomized to receive heparin 5000 U subcutaneous three times a day.
  Interventions: Drug: Heparin
- UFH 5000 U two times a day (Active Comparator): Study subjects will be randomized to receive heparin 5000 U subcutaneous two times a day.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin

SUMMARY:
This study is designed to assess: the incidence of abnormal partial thromboplastin time in patients receiving unfractionated heparin (UFH) 5000 U 2 times a day versus 3 times a day 72 hours after administration of the first dose of heparin.

Hypothesis: The basic hypothesis of this study is that patients receiving UFH 5000 U subcutaneously 3 times a day will have a higher proportion of elevated partial thromboplastin time than patients receiving UFH 5000 U subcutaneously twice a day.

DETAILED DESCRIPTION:
Administration of subcutaneous UFH for antithrombotic prophylaxis is standard therapy in the postoperative setting. Often, a dosage of 5000 U twice a day has been used, with a demonstrated antithrombotic efficacy and an acceptable hemorrhagic complication profile. However, recent surgery guidelines regarding antithrombotic prophylaxis with UFH 5000 U suggest that a thrice daily regimen should be used following major oncologic surgeries. These new guidelines have raised some concerns in anesthesiology, particularly regarding the safety of epidural catheters combined with thrice daily heparin. Optimal analgesia during the early postoperative period following some types of major oncologic surgery involves the placement of epidural catheters. Epidural analgesia provides the best relief of the significant pain which may be present after thoracotomy or supraumbilical laparotomy during the early postoperative period, improving ambulation, coughing, pulmonary function, bowel function as well as short and long-term quality of life. However, the benefits of epidural catheters must outweigh the risk of complications, the most feared being spinal hematoma. Recent guidelines in anesthesiology support the placement of epidural catheters with the concomitant administration of UFH 5000 U two times a day. However, these guidelines do not clearly support the placement of an epidural catheter if a three times a day regimen is used, very little data being available to assess the risk of this practice. Older studies (1973) suggest that a significant proportion of patients (15%) will develop abnormal partial thromboplastin times using a three times a day regimen. However, it is not known if these results are still consistent with more recent laboratory technologies, or how they compare to twice daily heparin. In the absence of even basic data regarding systemic effect on coagulation, it is difficult at this time to begin to determine safe practice regarding the placement of an epidural catheter in presence of a three times a day UFH 5000 U regimen. A recent pilot study conducted in our center showed that 20% (4/20) of patients receiving the thrice daily regimen will develop abnormal partial thromboplastin times at 72 hours following the first dose compared to 5% (1/20) in patients receiving the twice a day regimen. This larger scale study is designed to establish the incidence of abnormalities in partial thromboplastin times 72 hours following the administration of the first dose of heparin for both regimens.

Methods: 130 patients will be enrolled and divided in two equal groups (Group 1: to receive UFH 5000 U subcutaneous two times a day or Group 2: to receive UFH 5000 U subcutaneous three times a day)

As needed for standard anesthesia, surgical and post-operative care, an arterial line will be placed. Immediately prior the first UFH dose, a blood sample for partial thromboplastin time will collected through the arterial line. Since nutritional status may affect the patient's coagulation a blood sample to measure albumin and transthyretin will be collected simultaneously. The first dose of UFH will be given in the operating room by the anesthesiologist.

A second blood sample will be collected by venipuncture at 72 hours following the administration of the first dose of heparin.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective surgery by thoracoscopy requiring antithrombotic prophylaxis
* Anticipated duration of hospital stay of at least 3 days

Exclusion Criteria:

* Pre-existing coagulopathy
* Severe renal failure
* Known allergy to heparin
* History of heparin induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of abnormal partial thromboplastin time values 72 hours after the administration of the first dose of antithrombotic prophylaxis in patients receiving UFH 5000 U 2 times a day versus 3 times a day following surgery. | 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada